CLINICAL TRIAL: NCT06382506
Title: Can Hazelnut Flour Added to Gluten-free Corn Flour in Different Amounts Cause Differences in Blood Glucose Fluctuations?
Brief Title: The Effect of Hazelnut Flour on Blood Glucose
Acronym: Hazelnut
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Fatih Cesur, Assistant Professor, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024/138
Record Dates: First submitted 2024-02-17; First posted 2024-04-24 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Obesity; Celiac Disease; Blood Glucose; Flour Sensitivity
Keywords: Obesity; Celiac Disease; Blood glucose; Flour Sensitivity
MeSH Terms: conditions — Obesity; Celiac Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effect of cornbread consumption blood glucose fluctuations in participants. (Experimental): The bread contained 50 grams of digestible carbohydrates. Participants consumed these loaves of bread when they were hungry. Blood glucose measurements were taken at 0 (fasting),15, 30, 45, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Consumption of Cornbread with Hazelnut Bread
- The effect of cornbread with hazelnut bread consumption blood glucose fluctuations in participants. (Experimental): The bread contained 50 grams of digestible carbohydrates. Participants consumed these loaves of bread when they were hungry. Blood glucose measurements were taken at 0 (fasting),15, 30, 45, 60, 90, and 120 minutes.
  Interventions: Dietary Supplement: Consumption of Cornbread with Hazelnut Bread

INTERVENTIONS:
Dietary Supplement: Consumption of Cornbread with Hazelnut Bread — Cornbread was added to 15 grams and 30 grams of bread and consumed by the participants. Blood glucose levels were then measured. Obese and normal-weight individuals will be divided into two groups according to their anthropometric measurements.

SUMMARY:
One of the factors affecting human health is nutrition. The effects of foods on blood glucose are still under investigation. The Glycemic Index (GI), which is associated with many diseases today, is a value that measures the rate at which carbohydrate-containing foods raise blood glucose. It is thought that the loaves of bread produced will be a product with low GI value and can be consumed by celiacs and diabetics. It is aimed to investigate the effect of adding different amounts of hazelnut flour to bread recipes using gluten-free corn flour on blood glucose.

ELIGIBILITY:
Inclusion Criteria:

* The study group consisted of volunteer individuals aged between 18 and 35 years.
* The first blood glucose measurement was taken after at least 8 hours of fasting and any of the bread types were given to the participants for consumption.
* During the measurements, the volunteers were observed to avoid water, coffee, and any food intake and to avoid excessive exercise.

Exclusion Criteria:

* Pregnant,
* lactating women
* patients with physician-diagnosed chronic diseases

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-04-21 (Actual); Study Completion 2024-04-21 (Actual)

PRIMARY OUTCOMES:
One loaf of bread was consumed each week and the study will continue for a month. Blood glucose measurements were performed with a glucometer at 0 (fasting), 15, 30, 45, 60, 90, and 120 minutes after each bread consumption. | Within research completion, an average of a month
  The effect of loaves of bread with a high glycemic index on blood glucose is well known. The higher the glycemic index, the higher the blood glucose fluctuation. Glycemic index values should be lower than white bread. Consumption of hazelnut flour rich in fatty acids and fiber should show a positive change in blood glucose.

SECONDARY OUTCOMES:
This classification as obese and normal-weight individuals was made with the BIA (Bioelectrical impedance analysis) method. This classification was understood by anthropometric measurements made in the first week. | Within research completion, an average of 1 week
  It is known that high glycemic index values of bread consumption are paralleled by high blood fluctuations. On the other hand, the impact of bread consumption on obesity and normal-weight people is also of interest. In obese people, the high glycemic index predisposes them to overeating. As the amount of hazelnut flour in bread increases, there is a positive change in blood glucose fluctuations in individuals.

CONTACTS AND LOCATIONS:
Locations (1):
- Avrasya University, Trabzon, Turkey (Türkiye)

REFERENCES:
- [Derived] Cesur F, Uygur B. Can hazelnut flour added to gluten-free corn flour in different amounts cause differences in blood glucose fluctuations? Int J Food Sci Nutr. 2025 Feb;76(1):84-92. doi: 10.1080/09637486.2024.2435841. Epub 2024 Dec 3. PMID 39627012